CLINICAL TRIAL: NCT07348120
Title: Efficacy and Safety of Millet Seed Extract in the Treatment of Telogen Effluvium in Female Patients: A Randomized, Double-Blind, Controlled Trial
Brief Title: Efficacy and Safety of Millet Seed Extract in Telogen Effluvium Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, heba ahmed abdelgayed ibrahim, Lecturer of Dermatology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-95-2025
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Telogen Effluvium
Keywords: hair loss; millet seed extract; hair growth; biotin; telogen effluvium
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Millet Seed Extract Group (Experimental): Participants in this group received Millet seed extract capsules containing 420 mg millet seed extract, 200mcg biotin, 6mg L-cystine, and 27.48 mg vitamin B5, taken orally twice daily for 12 weeks.
  Interventions: Dietary Supplement: Millet Seed Extract group
- Control Group (Active Comparator): Participants in this group received capsules containing 5mg of biotin once daily for 12 weeks.
  Interventions: Dietary Supplement: Biotin group

INTERVENTIONS:
Dietary Supplement: Millet Seed Extract group — Millet seed extract capsules containing 420 mg millet seed extract, 200 mcg biotin, 6 mg L-cystine, and 27.48 mg vitamin B5, taken orally twice daily for 12 weeks. The extract is standardized to miliacin content.
  Arms: Millet Seed Extract Group
Dietary Supplement: Biotin group — Capsules containing 5 mg of biotin, taken orally once daily for 12 weeks.
  Arms: Control Group

SUMMARY:
This is a randomized, double-blind, controlled clinical trial investigating the efficacy and safety of millet seed extract capsules in treating telogen effluvium in female patients. The study will recruit 60 female participants with telogen effluvium who will be randomly assigned to receive either millet seed extract capsules (containing 420 mg millet seed extract, 200 mcg biotin, 6 mg L-cystine, and 27.48 mg vitamin B5) twice daily or Biotin forte capsules (5 mg biotin) once daily for 12 weeks. The primary outcome will measure changes in telogen and anagen hair densities using dermoscopy-assisted phototrichography. Secondary outcomes will assess patient satisfaction and unwanted body hair growth. Safety will be monitored throughout the study period at Cairo University's dermatology clinic.

DETAILED DESCRIPTION:
Telogen effluvium is characterized by diffuse hair shedding that significantly impacts quality of life. Millet seed extract, rich in bioactive compounds including miliacin, offers a promising natural treatment approach. This 12-week randomized, double-blind, controlled trial will recruit 60 female patients with telogen effluvium at Kasr Al Ainy, Cairo University. Participants will be randomly assigned to receive either millet seed extract capsules (420 mg millet seed extract, 200 mcg biotin, 6 mg L-cystine, 27.48 mg vitamin B5 twice daily) or biotin forte capsules (5 mg once daily). Primary outcome measures include telogen and anagen hair densities assessed by dermoscopy-assisted phototrichography at baseline and week 12. Secondary outcomes include patient satisfaction, unwanted body hair growth assessment, and Dermatology Life Quality Index scores. Safety will be monitored throughout the study period with adverse event reporting. The study includes female patients aged 18+ with clinically and trichoscopically confirmed telogen effluvium and hair shedding degree of 4 or higher on the Sinclair scale, excluding those with pregnancy, scalp diseases, or medication-induced hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Hair shedding degree of 4 or higher according to the Hair Shedding Visual Scale (Sinclair scale).
* Diagnosis of telogen effluvium confirmed by a dermatologist after ruling out other causes of non-scarring alopecia (e.g., alopecia areata, androgenetic alopecia).
* No use of topical or systemic hair loss treatments or oral hair growth supplements for at least 1 month prior to the study.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* History of scalp diseases or conditions affecting hair growth like androgenic alopecia and alopecia areata.
* Use of medications known to cause hair loss.
* Any underlying medical condition that could interfere with the study.
* Use of topical treatment in the last 3 month.
* Use of systemic treatment in the last 3 month such as iron, biotin or any hair growth supplements.
* Annemia or low serum level of ferritin.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Telogen and Anagen Hair Densities measured by Dermoscopy-Assisted Phototrichogram | Baseline (Week 0) and Week 12 of treatment
  Percentage change in telogen and anagen hair densities in the specified scalp area (external occipital protuberance region, 1.5 cm²) from baseline to week 12. Telogen and anagen densities will be calculated as the number of telogen/anagen hairs divided by total hair count in the selected area multiplied by 100. Measurements will be performed using dermoscopy-assisted phototrichogram (PTG) analysis with microphotographs taken on day 0 and day 7 of each assessment period

SECONDARY OUTCOMES:
Patient Satisfaction with Treatment using Visual Analogue Scale (VAS) | Week 12 (End of Study)
  Patient satisfaction will be measured using a 10-point visual analogue scale (VAS) where 0 = "Not satisfied at all" and 10 = "Completely satisfied". This assessment will be conducted at the end of the study (Week 12) to evaluate overall treatment satisfaction.
Unwanted Body Hair Growth Assessment | Baseline (Week 0) and Week 12 of treatment
  Clinical evaluation and dermoscopy-assisted phototrichogram analysis of unwanted body hair growth in a 4 cm x 4 cm standardized area on the anterior surface of the mid-thigh. Assessment includes visual macrophotograph evaluation for hair growth and density, and dermoscopic analysis using the same dermoscopy-assisted phototrichogram (PTG) technique applied to the scalp assessment.
Physician Global Assessment of Hair Improvement using Standardized Macrophotographs | Baseline (Week 0) and Week 12 (End of Study)
  Assessment of overall hair improvement by two blinded dermatologists and one non-blinded dermatologist using standardized macrophotographs taken at baseline and end of therapy. Scoring will use a 5-point scale: -1 = Worsening; 0 = No improvement; 1 = Mild improvement; 2 = Moderate improvement; 3 = Excellent improvement.
Patient Global Assessment of Overall Hair Improvement | Week 12 (End of Study)
  Patient self-assessment of overall hair improvement at the end of the study period using a 5-point scale: -1 = Worsening; 0 = No improvement; 1 = Mild improvement; 2 = Moderate improvement; 3 = Excellent improvement.
Change in Dermatology Life Quality Index (DLQI) Score | Baseline (Week 0) and Week 12 (End of Study)
  Assessment of the impact of telogen effluvium on quality of life using the validated Dermatology Life Quality Index (DLQI) questionnaire. The DLQI measures the effect of skin disease on patients' quality of life across six domains. Change from baseline to end of study will be evaluated.
Safety and Tolerability of Millet Seed Extract and Biotin Forte Capsules | Throughout the 12-week treatment period at Baseline (Week 0), Week 6, and Week 12
  Clinical evaluation and monitoring for any adverse effects including gastrointestinal discomfort, allergic reactions, and unwanted body hair growth. Adverse events will be graded for severity and documented including date of onset, duration, severity, action taken, and outcome. Serious adverse events will be reported to the principal investigator and ethics committee.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Aini Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center study with a small sample size, and de-identification cannot be fully guaranteed. Aggregate results, including summary statistics and outcome analyses, will be made available through publication